CLINICAL TRIAL: NCT02635971
Title: A Randomized Controlled Phase II Study on Intra-arterial Versus Intravenous Chemotherapy Infusion With Gemcitabine and Oxaliplatin for Locally Advanced Pancreatic Cancer
Brief Title: Intra-arterial Versus Intravenous Chemotherapy for Locally Advanced Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiqiang Meng, Professor, MD, Ph D, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAI-2015
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Carcinoma, Pancreatic
Keywords: transcatheter arterial infusion; randomized controlled trial; chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAI chemotherapy (Experimental): Patients in this arm will receive transcatheter arterial infusion of chemotherapy with gemcitabine and oxaliplatin every 2 weeks, until progression of disease or adverse effects leading to treatment termination. Each 4-week period is one cycle of treatment.
  Interventions: Procedure: Transcatheter arterial infusion; Drug: Gemcitabine; Drug: Oxaliplatin
- Chemotherapy (Active Comparator): Patients in this arm will receive intravenous chemotherapy with gemcitabine and oxaliplatin every 2 weeks, until progression of disease or adverse effects leading to treatment termination. Each 4-week period is one cycle of treatment.
  Interventions: Procedure: Intravenous chemotherapy; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Procedure: Transcatheter arterial infusion
  Arms: TAI chemotherapy
Procedure: Intravenous chemotherapy
  Arms: Chemotherapy
Drug: Gemcitabine
Drug: Oxaliplatin

SUMMARY:
This study aims to explore the efficacy and safety of intra- arterial infusion of gemcitabine and oxaliplatin in locally advanced pancreatic cancer. This protocol is overseen by the Fudan University Institutional Review Board which has Federal Wide Assurance through the U.S. Department of Health & Human Services (Approved: April 25, 2002).

DETAILED DESCRIPTION:
Primary Outcome Measures:

To compare the overall survival (OS) in patients with locally advanced pancreatic cancer treated with transcatheter arterial infusion (TAI) of chemotherapeutics or systemic delivered chemotherapy.

Secondary Outcome Measures:

To compare the progression free survival (PFS), objective response rate (ORR), quality of life (QoL), and adverse effects of treating locally advanced pancreatic cancer patients with TAI or systemic chemotherapy.

Exploratory Outcome Measures:

To evaluate the correlation between prognosis and expression of serum microRNAs of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed unresectable locally advanced pancreatic adenocarcinoma.
* Measurable disease by RECIST criteria must be present.
* Karnofsky Performance Status ≥ 70
* Patients with adequate organ functions reflected by the laboratory criteria below:

Granulocytes ≥ 1,500/uL Hemoglobin ≥ 8.0 gm/dL Platelets ≥ 100,000/uL Serum creatinine < 2.0 mg/dL Bilirubin < 1.5 mg/dL SGPT < 2.5 x normal Alk Phos < 2.5 x normal

* Prior local therapy, e.g., radiation, is allowed provided that at least 4 weeks washout time is given.
* Patients with jaundice must have a biliary drainage decompression operation before recruitment.
* Patients must not be pregnant. Serum beta-HCG will be checked in all premenopausal patients.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Subject with metastatic disease.
* Prior treatment with systemic chemotherapy.
* Known allergies to the gemcitabine, oxaliplatin or iodine contrast agent.
* Subject with Child-Pugh grade Class C hepatic impairment, active gastrointestinal bleeding, severe coagulation disorder that could not be corrected，or other contraindication for transcatheter infusion.
* Untreated or uncontrolled deep vein thrombosis, arterial thrombosis of lower extremity, or aneurysm.
* Concurrent infection requiring intravenous antibiotics.
* Skin injury or infection of groin area, or other situation that not appropriate for femoral artery puncture.
* Other serious illness or condition including cardiac disease including congestive heart failure (New York Heart Association Classification III or IV), active HIV infection/HIV disease, psychiatric disorders.
* Known central nervous system involvement and leptomeningeal disease
* Subject with previous or concurrent cancer that is distinct in primary site or histology from pancreatic adenocarcinoma except cervical carcinoma in situ, non-melanoma carcinoma of the skin or in situ carcinoma of the bladder. Any cancer curatively treated greater than 3 years prior to entry is permitted.
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death, assessed up to 100 months.

SECONDARY OUTCOMES:
Progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Meng, MD, Ph D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang C, Cheng CS, Shen Y, Chen H, Lin J, Hua Y, Feng L, Wu C, Wang P, Chen Z, Meng Z. Digital subtraction angiography-guided pancreatic arterial infusion of GEMOX chemotherapy in advanced pancreatic adenocarcinoma: a phase II, open-label, randomized controlled trial comparing with intravenous chemotherapy. BMC Cancer. 2024 Aug 2;24(1):941. doi: 10.1186/s12885-024-12695-8. PMID 39095759